CLINICAL TRIAL: NCT04900441
Title: Determination of Long Term Rehabilitation Needs and Assessment of Functional Capacity in Individuals With COVID-19 With Tele-assessment Methods
Brief Title: Tele-assessment in Individuals With COVID-19
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Gulhan Yilmaz Gokmen, Assistant Professor, Bandırma Onyedi Eylül University
Other Study IDs: GYGokmen
Record Dates: First submitted 2021-05-21; First posted 2021-05-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: COVID-19; tele-assessment; C19-YRS; rehabilitation needs; functional capacity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In most countries, after the measures taken to reduce the effects of the epidemic and quarantine practices, a remote screening tool has emerged in order to screen the needs developing after COVID-19 and to make the necessary rehabilitation applications in time. Sivan et al. A comprehensive multi-system phone scan of the COVID-19 Yorkshire Rehabilitation Screening Tool (C19-YRS) has been developed by a multidisciplinary rehabilitation team.

This study, which will be carried out using the C19-YRS tool and the 30-second sit-and-go test that evaluates functional capacity and mobility conditions, is expected to contribute to the clinical and literature since most of the studies on COVID-19 focused only on the acute and subacute periods. In addition, considering the pandemic conditions all over the world, it will be possible to benefit from the advantages of the tele-assessment application and by reaching more people, possible clinical problems/needs and whether there is a change functional capacities in individuals after COVID-19 will be identified.

ELIGIBILITY:
Inclusion Criteria

* being 18 years of age or older,
* Patients who have had COVID-19 and whose treatment was completed and the PCR test was negative for 2 times or who passed the positive PCR test for 28 days,
* Individuals who can take and execute verbal orders,
* giving consent on a voluntary basis

Exclusion Criteria:

* individuals who have not had covid 19 or Acute-stage patients with COVID-19
* individuals who refuse to participate in the tele-assessment
* individuals with dementia, cognitive problems or communication problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had COVID-19 and whose treatment was completed and the PCR test was negative for 2 times or who passed the positive PCR test for 28 days
Sampling Method: Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Covid-19 Yorkshire Rehab Screen (C19YRS) | Baseline
  The C19YRS was developed as a screening tool to monitor long-term symptoms due to Covid-19. The screening tool covers 19 items which combines yes/no answers and an 11 point ordinal scale (0-10) where a higher score denotes increased symptom severity.
30-sec sit and go test | Baseline
  It will be used for functional evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz Gokmen G, Durmaz D, Demir C, Yilmaz FN. Determining Post-COVID-19 Symptoms and Rehabilitation Needs in Hospitalized and Nonhospitalized COVID-19 Survivors with Tele-Assessment Methods. Telemed J E Health. 2023 Sep;29(9):1312-1323. doi: 10.1089/tmj.2022.0349. Epub 2023 Feb 9. PMID 36757300